CLINICAL TRIAL: NCT05321849
Title: Echocardiography-guided Percutaneous Patent Ductus Arteriosus Closure: A One-Year Single Centre Experience in Indonesia
Brief Title: Echocardiography-guided Percutaneous Patent Ductus Arteriosus Closure
Status: Completed | Type: Observational
Sponsor: National Cardiovascular Center Harapan Kita Hospital Indonesia (Other)
Responsible Party: Principal Investigator, Sisca Natalia Siagian, Principal Investigator, National Cardiovascular Center Harapan Kita Hospital Indonesia
Other Study IDs: LB.02.01/VII/475/KEP076/
Record Dates: First submitted 2022-03-22; First posted 2022-04-11 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Echocardiography; PDA
Keywords: Patent Ductus Arteriosus (PDA); Transcatheter closure; Without fluoroscopy; echocardiography
MeSH Terms: conditions — Ductus Arteriosus, Patent

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Use Fluoroscopy (Control): PDA closure in 30 patients with fluoroscopy guide
- No fluoroscopy (test): PDA closure in 30 patients with echocardiography guide, without fluoroscopy
  Interventions: Other: Echocardiography guide

INTERVENTIONS:
Other: Echocardiography guide — Patients with PDA are percutaneously closed with echocardiography guide, without fluoroscopy like classical procedures
  Groups: No fluoroscopy (test)

SUMMARY:
Since the first successful percutaneous closure under transoesophageal echocardiographic (TEE) guidance, many centres explored transcatheter procedures without fluoroscopy. This single centre study aims to show the feasibility and safety of percutaneous patent ductus arteriosus (PDA) closure under echocardiography-only guidance during our one-year experience. Patients with PDA were recruited for percutaneous PDA closure guided by either fluoroscopy or echocardiography-only in National Cardiovascular Center Harapan Kita. Patients were evaluated clinically and radiologically using TTE at 6, 24 and 48 hours after the procedure. Primary endpoint was the procedural success. Secondary endpoints were the procedural time and the rate of adverse events. Echocardiography-guided PDA closure is non-inferior to fluoroscopy-guided PDA closure, with similar procedural times. However, this method is operator-dependent and requires an experienced team for it to be performed successfully.

DETAILED DESCRIPTION:
From March 2019 to April 2020, a total of 60 patients with PDA were recruited as participants for this prospective, single-centre, non-randomized clinical trial. They were divided equally into two groups: the fluoroscopy group who underwent percutaneous PDA guided by fluoroscopy and the echocardiography group who underwent percutaneous PDA closures guided by transthoracic echocardiography (TTE) and TEE at the National Cardiovascular Centre Harapan Kita, Jakarta, Indonesia. Patients with stable hemodynamic and clinically asymptomatic PDA were evaluated and considered for transcatheter PDA closure. Significant chamber enlargement and mild to moderate pulmonary hypertension were also indications for transcatheter closure. Ductal morphology was evaluated using multiplanar TTE and TEE imaging.

After the procedures, patients were evaluated and followed-up after 6, 24 and 48 hours to observe any residual shunts and complications. This study protocol conforms to the ethical guidelines of the Declaration of Helsinki and the Nuremberg Code with approval from the Research Ethics Committee of National Cardiovascular Center Harapan Kita No LB.02.01/VII/475/KEP076/2020. Written consent to perform the procedure and to use the patients' medical records for this study was obtained from the patients or their parents.

ELIGIBILITY:
Inclusion Criteria:

* PDA, age <= 18yo

Exclusion Criteria:

* >= 18yo, Eisenmenger syndrome, coexistence of other associated congenital heart disease

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The inclusion criteria for this study are children under 18 years old with PDA who were planned for PDA closure. The exclusion criteria include the coexistence of other associated congenital heart disease requiring surgical intervention and PDA patients with irreversible high pulmonary vascular resistance (PVR) unreactive with the oxygen test.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-03-12 (Actual); Primary Completion 2020-06-23 (Actual); Study Completion 2020-06-23 (Actual)

PRIMARY OUTCOMES:
Change of Residual Shunt from post-procedure to 6 hours, 24 hours and 48 hours | 6, 24 hours, and 48 hours
  PDA residual shunt post PDA closure
Change of Device Position from post-procedure to 6 hours, 24 hours and 48 hours | 6, 24 hours, and 48 hours
  If device dislodge during follow-up

SECONDARY OUTCOMES:
Procedural time | 6hours
  Time total needed to complete procedure
Complication | 6, 24hours, and 48hours
  if any death, peripheral vascular injury, pericardial effusion, pericardial tamponade

CONTACTS AND LOCATIONS:
Overall Officials: Sisca N Siagian, MD, Principal Investigator — National CCHK
Locations (1):
- National Cardiovascular Center Harapan Kita Jakarta Indonesia, Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No
At the moment, we have no plan to share the whole participant data. However, if it is needed, we will.

REFERENCES:
- [Derived] Siagian SN, Prakoso R, Putra BE, Kurniawati Y, Lelya O, Sembiring AA, Atmosudigdo IS, Roebiono PS, Rahajoe AU, Harimurti GM, Mendel B, Christianto C, Setiawan M, Lilyasari O. Echocardiography-Guided Percutaneous Patent Ductus Arteriosus Closure: 1-Year Single Center Experience in Indonesia. Front Cardiovasc Med. 2022 May 23;9:885140. doi: 10.3389/fcvm.2022.885140. eCollection 2022. PMID 35677684